CLINICAL TRIAL: NCT05892328
Title: Dose Response Effect of Watermelon Consumption on Ambulatory Blood Pressure in Adults With Pre-hypertension: A Randomized Controlled Pilot Trial
Brief Title: Watermelon Dose Response Blood Pressure Study
Acronym: WMBP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: National Watermelon Promotion Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-2023-03
Record Dates: First submitted 2023-05-02; First posted 2023-06-07 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Pre-hypertension; Cardiovascular Diseases
Keywords: Watermelon; Blood pressure; Pre-hypertension
MeSH Terms: conditions — Prehypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The proposed trial will be a randomized, 3 arm, placebo-controlled, parallel study design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Calorie-matched control beverage
  Interventions: Other: Control
- Watermelon flesh Dose 1 (Active Comparator): 1 cup watermelon flesh, ~152 g
  Interventions: Other: Watermelon Flesh Dose 1
- Watermelon flesh Dose 2 (Active Comparator): 2 cups watermelon flesh, ~304 g
  Interventions: Other: Watermelon Flesh Dose 2

INTERVENTIONS:
Other: Watermelon Flesh Dose 1 — 1 cup watermelon flesh, ~152g, 7 days/week over a 4-week period
  Arms: Watermelon flesh Dose 1
Other: Watermelon Flesh Dose 2 — 2 cups watermelon flesh, ~304 g, 7 days/week over a 4-week period
  Arms: Watermelon flesh Dose 2
Other: Control — 304g italian ice, 0 g watermelon, 7 days/week over a 4-week period
  Arms: Control

SUMMARY:
1. Primary outcome: To evaluate the dose response effects of watermelon flesh in regulating Blood Pressure (BP) in individuals with pre-hypertension.
2. Secondary outcomes: To study the dose-response effects of watermelon flesh intake on cardio-metabolic risk factors including plasma metabolic markers, lipid profile and nitrate/nitrite levels in individuals with pre-hypertension.

DETAILED DESCRIPTION:
The proposed study will be conducted in humans according to Good Clinical Practice (GCP) guidelines. All subjects will review and sign an Informed Consent Form approved by the Illinois Institute of Technology's Institutional Review Boards (IRB) prior to screening.

The proposed study is a randomized, three-arm (n=12/arm), single-blinded, placebo-controlled, 4-week, parallel study design in individuals with pre-hypertension (systolic BP ≥ 120-139 mm Hg or a diastolic BP ≥ 80-89 mm Hg).

Pre-Screening: To learn more about the study and to pre-qualify, potential subjects can call the Clinical Nutrition Research Center (CNRC) or visit the website posted on recruitment flyers or from other recruitment materials. If individuals call the CNRC, a staff member will provide a brief background on the study and ask a series of questions from a pre-screening questionnaire to assess eligibility. The same questionnaire is available on the website and can be filled out by potential subjects online. The pre-screening questionnaire includes self-reported information about health status and lifestyle factors that can be used to determine if someone is not eligible for the study.

Screening: Participants will be asked to read, ask questions, sign and date the Institutional Review Board (IRB) approved Informed Consent Form (ICF) before any laboratory or study screening procedures begin. Participants will be informed of study procedures and schedules. Once ICF is signed by participant and staff, height, weight and waist circumference measurements, vital signs measurements, body temperature measurements (by contactless thermometer), and a finger prick (to confirm fasting status and blood sugar) will be collected.

Pre-Study Visit: If participants are eligible and willing to continue, a pre-study visit will be scheduled. The pre-study visit is for training on various aspects of the study. Participants will have diet counseling on foods that are rich in the components typically found in watermelon (e.g. tomatoes, carrots, sweet potatoes, etc.). Participants will be asked to avoid these foods for at least 7 days before the first study visit day. There will also be coaching on how to complete a 3-day food record that will be collected at each study visit.

At the Pre-Study Visit study participants will be randomized equally to each test group (n=12/group) according to a computer-generated randomization sequence. Participants will receive one of the three study test beverages:

1. Control (0 g watermelon),
2. Watermelon flesh Dose 1 (WF1, 1 cup watermelon flesh, ~152 g) or
3. Watermelon flesh Dose 2 (WF2, 2 cups watermelon flesh, ~304 g);

Study Visit Days: There will be 3 study days that will take approximately 1-1.5 hours. Study visit days will occur on day 0, 14, and 30. Before each study visit participants will be asked to consume a fixed dinner the night before at least 10 hours prior to the visit. A 3-day food record will be collected at the visit.

Measurements include height, weight, waist circumferences, blood pressure, body temperature, heart rate, and fasting blood glucose. A fasting urine and blood sample will then be collected.

Participants will consume the first study test beverage (Control, WF1 or WF2) on-site and will be given test beverages to take home and instructed to consume the beverage every day in the morning between 8-10 am for 4 weeks. Treatment beverages will be given to the participant to consume over the next 2 weeks at day 14 (visit 3). 24-hour Ambulatory Blood Pressure Machine (ABPM) will be distributed after consuming the test beverages on day 0 and day 28 during the visit.

Follow up visits: 24-hours after visit 1 and 4, ABPM machines will be returned. Treatment beverages will be given to the participant to consume over the next 2 weeks at the first follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are nonsmokers
* Healthy overweight/ obese man or woman between 25 and 65 years of age
* Blood pressure 120-160 mmHg systolic or 80-100 mm/Hg diastolic at screening visit
* Fasting blood glucose concentration between 100 mg/dL and 125 mg/dL at screening visit (value range indicate prediabetes, by finger prick and/or venous blood sampling)
* Have no clinical evidence/history of cardiovascular, metabolic, respiratory, renal, gastrointestinal, or hepatic disease

Exclusion Criteria:

* Smoker
* Vegetarian
* Men and women who have fasting blood glucose concentration <100 or >125 mg/dL at screening visit
* Uncontrolled blood pressure ≥140 mmHg (systolic)/ ≥ 90 mmHg (diastolic)
* Over the counter supplements (e.g. fiber supplements, probiotics and/or prebiotics, antioxidants, anti-inflammation)
* Dietary supplements like (garlic, fish oil), glutamine supplements, grape seed extract, L-citrulline/arginine
* Cholesterol-lowering medications, anticoagulants, blood pressure-lowering medications,) and/or taking prescription medications that may interfere with study procedures or endpoints (e.g. gastrointestinal medications, antibiotics) within the last 30 days
* Have cancer other than non-melanoma skin cancer in previous 5 years
* Taking unstable dose of hormonal contraceptive and/or a stable dose less than 6 months
* Planning to become pregnant, pregnant and/or breast-feeding
* Excessive exerciser or a trained athlete
* Drink excessive amount of coffee/tea (> 5 cups per day)
* Donated blood within last 3 months
* Have allergies/intolerances to foods consumed in the study
* Currently eat > 2 servings of watermelons per day
* Actively losing weight/ trying to lose weight (unstable body weight fluctuations of > 11 lbs in 3 months)
* Addicted to drugs or alcohol
* Have significant psychiatric or neurological disturbances that may interfere with the ability to follow the study protocol

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the change in the dose response effects of watermelon flesh in regulating BP in individuals with pre-hypertension. | Baseline to 4 weeks
  This objective will be accomplished by assessing the 24-h Ambulatory Blood Pressure Machine (ABPM) in individuals with pre-hypertension before and after 4 weeks of watermelon flesh intake. Two doses of watermelon flesh will be tested (1 and 2 cup servings) compared to control.

SECONDARY OUTCOMES:
To evaluate the change in lipid profile in individuals with pre-hypertension after consuming watermelon flesh. | Baseline to 4 weeks
  Randox automated clinical analyzer measuring total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides
To evaluate the change in plasma and urine nitrite/nitrate in individuals with pre-hypertension after consuming watermelon flesh. | Baseline to 4 weeks
  Plasma and urine nitrate ad nitrite concentrations will be measured using Griess assay
To evaluate the change in glucose in individuals with pre-hypertension after consuming watermelon flesh. | Baseline to 4 weeks
  Randox automated clinical analyzer measuring glucose
To evaluate the change in insulin in individuals with pre-hypertension after consuming watermelon flesh. | Baseline to 4 weeks
  Randox automated clinical analyzer measuring glucose
To evaluate the changes in L-Citrulline, Arginine, and Asymmetric Dimethylarginine (ADMA) in individuals with pre-hypertension after consuming watermelon flesh, analyzed by mass spectrometry. | Baseline to 4 weeks
  Collected plasma samples will be extracted with 0.1% formic acid in isopropanol. The samples will be centrifuged, filtered and analyzed for L-citrulline, arginine and ADMA on ultra-high performance liquid chromatography triple quadrupole mass spectrometry (UHPLC-QQQ-MS)

CONTACTS AND LOCATIONS:
Overall Officials: Indika Edirisinghe, Ph.D., Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States